CLINICAL TRIAL: NCT06199596
Title: The Effect of Alpha-s1 Casein Hydrolysate for Patients With Chronic Insomnia: A Randomized Double-Blind Controlled Trial
Brief Title: Alpha-s1 Casein Hydrolysate on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Chief, Department of Neurology Affiliation: Kuang Tien General Hospital, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KTGH11008
Record Dates: First submitted 2023-12-15; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Chronic Insomnia; Polysomnography
Keywords: Alpha-s1 casein hydrolysate; Randomized controlled trial; insomnia; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACH (Aalpha-s1 casein hydrolysate) (Experimental): Each participant will take Prelactium capsules (alpha-s2 casein hydrolysate supplement; 150mg per capsule) 30 minutes before bedtime for a duration of 4 weeks: 4 capsules in the first two weeks and 2 capsules in the last two weeks.
  Interventions: Dietary Supplement: alpha-s1 casein hydrolysate
- Placebo (Maltodextrin) (Placebo Comparator): Each participant will take Maltodextrin capsules (150mg per capsule) 30 minutes before bedtime for a duration of 4 weeks: 4 capsules in the first two weeks and 2 capsules in the last two weeks.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: alpha-s1 casein hydrolysate — 150mg of Prelactium per capsule
  Other Names: Prelactium
  Arms: ACH (Aalpha-s1 casein hydrolysate)
Dietary Supplement: Maltodextrin — 150mg of Maltodextrin per capsule
  Arms: Placebo (Maltodextrin)

SUMMARY:
This study investigates the impact of Aalpha-s1 casein hydrolysate (ACH; Lactium®) on sleep quality in individuals with chronic insomnia, employing both subjective sleep profiles and objective polysomnography (PSG) recordings.

DETAILED DESCRIPTION:
During the trial, the use of food or health products containing sedative or hypnotic ingredients or formulations is prohibited.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 80 who meet the diagnostic criteria for chronic insomnia according to the International Classification of Sleep Disorders (ICSD) (Third Edition);
2. PSQI score greater than 5;
3. participants must voluntarily agree to participate in the trial after explanation by a physician and complete the informed consent form.

Exclusion Criteria:

1. currently using tranquilizers, hypnotics, or stimulant-related medications or substances (such as coffee or energy drinks);
2. patients with a history of significant head trauma;
3. individuals with alcohol abuse within the past year;
4. those with other severe medical conditions (e.g., hepatic or renal dysfunction);
5. Pregnant women or breastfeeding mothers;
6. participants unable to comply with the trial schedule;
7. individuals on a vegetarian diet;
8. those with allergies to dairy products.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 2nd and 4th week
  A sleep-related questionnaire, ranging from 0 to 28, where higher scores indicate more acute symptoms of insomnia.
Pittsburgh Sleep Quality Index (PSQI) | 2nd and 4th week
  A sleep-related questionnaire, ranging from 0 to 21 with the higher total score indicating worse sleep quality.
Epworth Sleepiness Scale (ESS) | 2nd and 4th week
  A sleep-related questionnaire, ranging from 0 to 24. Scores from 0 to 10 reflect normal levels of daytime sleepiness, and scores over 10 are considered to reflect excessive daytime sleepiness.
General Sleep Disturbance Scale (GSDS) | 2nd and 4th week
  A sleep-related questionnaire, ranging from 0 (no disturbance) to 147 (extreme sleep disturbance).
Hospital Anxiety and Depression Scale (HADS) | 2nd and 4th week
  A sleep-related questionnaire, ranging from 0 to 21. A total score of >8 points denotes considerable symptoms of anxiety or depression.
Sleep quality | baseline and 4th week
  Polysomnography (PSG)

CONTACTS AND LOCATIONS:
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan